CLINICAL TRIAL: NCT04828057
Title: Preservative-free Fixed-dose Combination of Tafluprost 0.0015% / Timolol 0.5% in Patients With Open-angle Glaucoma or Ocular Hypertension: Clinical Effectiveness, Tolerability and Safety in a Real World Setting
Status: Completed | Type: Observational
Sponsor: Santen Pharmaceutical (Taiwan) Co., LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: TW-VISIONARY Study
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Ocular Surface Disease; Primary Open Angle Glaucoma
Keywords: tafluprost; Tapcom-s; switching
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — tafluprost; Timolol; Latanoprost; Bimatoprost; Travoprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tafluprost, timolol maleate — Patients prescribe PG mono who occurs OSD or I IOP lower insufficient. patients switch to combination therapy.
  Other Names: latanoprost; tafluprost; bimatoprost; travoprost

SUMMARY:
The primary objective of this study is to assess the effectiveness of Tafluprost / Timolol in controlling ocular hypertension, as measured by mean change in intra-ocular pressure (IOP) from baseline to after 6 months of treatment from initiation, in patients with open angle glaucoma (OAG) or ocular hypertension (OHT), who do not respond sufficiently to initial topical treatment, in routine clinical practice.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effectiveness of Tafluprost / Timolol in controlling ocular hypertension, as measured by mean change in intra-ocular pressure (IOP) from baseline to after 6 months of treatment from initiation, in patients with open angle glaucoma (OAG) or ocular hypertension (OHT), who do not respond sufficiently to initial topical treatment, in routine clinical practice.

This study will include adults with open angle glaucoma or ocular hypertension, who received their first Tafluprost / Timolol prescription at baseline, even if Tafluprost / Timolol was not continued after the first prescription. In addition, patients must have their IOP recorded within 7 days before their first prescription of Tafluprost / Timolol, in order to be eligible for this study. Only those who provide informed consent will be included.

At the time of a scheduled clinic visit, eligible patients will be invited to participate in the study and willing patients will be requested to sign an informed consent form. Once informed consent is obtained, the patient is included in the study and relevant data will be recorded during routine clinical visits. Participation in this study is entirely voluntary; any patient may withdraw consent to participate in this study at any time. The withdrawn patient's data will not be analyzed in this study and the number of patients who withdrew consent will appear in the final study report.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study-related activities (study-related activities are any procedure related to extraction of data according to the protocol)
* According to the approved indications of Tafluprost / Timolol as indicated in the SPC

  * Male or female patients ≥20 years of age at time of informed consent
  * Diagnosis of open angle glaucoma or ocular hypertension
  * Insufficient IOP control with a monotherapy utilizing topical prostaglandin analogues, necessitating the use of a combination therapy according to the judgement of the treating ophthalmologist
  * Patient judged by their physician to benefit from preservative free eye drops
* Not used Tafluprost / Timolol before

Exclusion Criteria:

* Patient pregnant or nursing
* Pregnancy planned in the following 6 months
* Presence of contraindications as listed in the SPC
* Any ophthalmologic surgery within 6 months prior to the study
* Participation in any other investigational study within 30 days prior to enrolment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for the current study is all eligible patients who received at least one prescription of Tafluprost / Timolol in Taiwan; however, the sample population will be limited to eligible patients in the clinics included in the study
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Mean change of intraocular pressure (IOP) | 6 months post initiation
  The primary endpoint will be assessed for the whole patient group and separately in specific subgroups according to their last glaucoma treatments before initiating Tafluprost / Timolol. Classification of prior therapy

SECONDARY OUTCOMES:
Mean change in intra-ocular pressure (IOP) from baseline to after 4 and 12 weeks | from baseline to after 4 and 12 weeks of treatment from initiation
  Mean change in intra-ocular pressure (IOP) from baseline to after 4 and 12 weeks of treatment from initiation
Proportion of responders at 12 weeks, defined as change from baseline IOP of 20% or more | 12 weeks post initiation
  Proportion of responders at 12 weeks,defined as change from baseline IOP of 20% or more
Evaluation of clinical signs with Tafluprost / Timolol | 6 months post initiation
  o Change in conjunctival hyperaemia distribution by severity
Change in the evaluation of subjective symptoms with Tafluprost / Timolol. Difference in distribution by severity. Severity categorized as none, mild, moderate, severe. | 6 months post initiation
  o Dry eye
Evaluation of the effectiveness (IOP-development) of Tafluprost / Timolol by the physician as measured by change in distribution by severity | 6 months post initiation
  * Better than prior medication
  * Same as prior medication
  * Worse than prior medication
Evaluation of clinical signs during therapy with Tafluprost / Timolol by the physician as measured by change in distribution by severity | 6 months post initiation
  * Better than prior medication
  * Same as prior medication
  * Worse than prior medication
Evaluation of tolerability of Tafluprost / Timolol by the Patient as measured by change in distribution by severity | 6 months post initiation
  * Very good
  * Good
  * Satisfactorily
  * Poor
Physician assessment of patient compliance compared to previous therapy | 6 months post initiation
  * Better
  * Equal
  * Worse
Concomitant therapy for glaucoma | 6 months post initiation
  Record concomitant therapy from baseline to 6 months post initiation
Evaluation of clinical signs with Tafluprost / Timolol | 6 months post initiation
  o Change in corneal fluorescein staining (CFS) distribution by severity. Optional
Evaluation of clinical signs with Tafluprost / Timolol | 6 months post initiation
  o Mean change in Visual acuity (VA)
Evaluation of clinical signs with Tafluprost / Timolol | 6 months post initiation
  o Mean change in Schirmer's test. Optional
Evaluation of clinical signs with Tafluprost / Timolol | 6 months post initiation
  o Mean change in tear break up time (TBUT). Optional
Change in the evaluation of subjective symptoms with Tafluprost / Timolol. Difference in distribution by severity. Severity categorized as none, mild, moderate, severe. | 6 months post initiation
  o Irritation
Change in the evaluation of subjective symptoms with Tafluprost / Timolol. Difference in distribution by severity. Severity categorized as none, mild, moderate, severe. | 6 months post initiation
  o Itching eyes
Change in the evaluation of subjective symptoms with Tafluprost / Timolol. Difference in distribution by severity. Severity categorized as none, mild, moderate, severe. | 6 months post initiation
  o Foreign body sensation
Change in the evaluation of subjective symptoms with Tafluprost / Timolol. Difference in distribution by severity. Severity categorized as none, mild, moderate, severe. | 6 months post initiation
  o Eye pain
Change in the evaluation of subjective symptoms with Tafluprost / Timolol. Difference in distribution by severity. Severity categorized as none, mild, moderate, severe. | 6 months post initiation
  o Other

CONTACTS AND LOCATIONS:
Overall Officials: Wei-wen Su, Principal Investigator — Chang-Geng Medical Foundation Linkou Chang-Geng Memorial Hospital
Locations (1):
- Chang-Geng Medical Foundation Linkou Chang-Geng Memorial Hospital, Taoyuan, Taiwan